CLINICAL TRIAL: NCT00005631
Title: Cytoreduction and Stem Cell Mobilization With Rituximab and ICE for Patients With Refractory or Relapsed CD20+ B-Cell IGL Eligible for ASCT: The RICE Protocol
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Large Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-092; CDR0000067785 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1774
Record Dates: First submitted 2000-05-02; First posted 2004-02-16 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic | interventions — Filgrastim; Rituximab; Carboplatin; Etoposide; Ifosfamide

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: carboplatin
Drug: etoposide
Drug: ifosfamide

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining combination chemotherapy with monoclonal antibody therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab and combination chemotherapy in treating patients who have relapsed or refractory large cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete response rate in patients with relapsed or refractory CD20-positive diffuse large cell, immunoblastic, or anaplastic large cell lymphoma treated with cytoreduction and mobilization with rituximab, ifosfamide, carboplatin, and etoposide (RICE). II. Assess the ability of this regimen to deplete the stem cell harvest of B-cells and tumor cells in these patients. III. Assess the efficacy of this regimen to mobilize peripheral blood progenitor cells in these patients. IV. Assess the safety and toxicity of this regimen in these patients.

OUTLINE: Cytoreduction and mobilization: Patients receive ifosfamide IV over 24 hours and carboplatin IV on day 4 and etoposide IV over 1 hour on days 3-5. Chemotherapy repeats every 2 weeks for 3 courses. Patients receive rituximab IV on day -2 before initiation of chemotherapy and on day 1 of each course of chemotherapy. Patients receive filgrastim (G-CSF) subcutaneously (SC) daily on days 7-14 of each course of chemotherapy. Patients with complete or partial response after completion of course 3 continue to receive G-CSF SC daily until peripheral blood stem cells (PBSC) are harvested. When blood counts recover, PBSC are harvested and selected for CD34+ cells. If sufficient numbers of CD34+ cells are not obtained, patients undergo bone marrow harvest.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven non-Hodgkin's lymphoma that is in first relapse or refractory to primary therapy Eligible types: Diffuse large cell Immunoblastic Anaplastic large cell Eligible for autologous peripheral blood stem cell transplantation CD20-positive disease Measurable disease No brain parenchyma involvement

PATIENT CHARACTERISTICS: Age: 18 to 72 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 50,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL unless due to Gilbert's disease No chronic or persistent hepatitis Hepatitis B surface antigen negative Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min No chronic renal insufficiency Cardiovascular: Normal baseline cardiac function Ejection fraction at least 50% by echocardiogram or MUGA scan No myocardial infarction within the past 6 months No unstable angina No cardiac arrhythmias except chronic atrial fibrillation Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception HIV negative No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No uncontrolled infection

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Prior rituximab allowed Chemotherapy: No prior carboplatin or cisplatin Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Kewalramani T, Zelenetz AD, Nimer SD, Portlock C, Straus D, Noy A, O'Connor O, Filippa DA, Teruya-Feldstein J, Gencarelli A, Qin J, Waxman A, Yahalom J, Moskowitz CH. Rituximab and ICE as second-line therapy before autologous stem cell transplantation for relapsed or primary refractory diffuse large B-cell lymphoma. Blood. 2004 May 15;103(10):3684-8. doi: 10.1182/blood-2003-11-3911. Epub 2004 Jan 22. PMID 14739217